CLINICAL TRIAL: NCT06333288
Title: Pilot Trial to Evaluate PROblem Solving Therapy and APPLE Watch for College Students (PRO-APPLE)
Brief Title: Pilot Trial to Evaluate PROblem Solving Therapy and APPLE Watch for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Hagar Hallihan, Research Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0268
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: PRO-APPLE Study is a 2-arm pilot Randomized Control Trial (RCT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Other): The intervention group will receive individual PST (60 min individual sessions for 6 weeks, in addition to engaging with APPLE Watch features including fitness tracking (such as regular walks), heart rate, and sleep management on a daily basis. Throughout the final 6 individual self-engaged sessions, participants will persist in engaging and utilizing APPLE Watch features, incorporating daily fitness tracking (such as regular walks), wellness applications, and sleep management and apply PST.
  Interventions: Behavioral: PST-APPLE Watch group
- Control group (Other): Participants assigned to Education-only control will be asked to watch "Quit Drinking Motivation," a 20-min video created by the MotivationHub. This video consists of a speech and conversation discussing the negative consequences resulting from their alcohol misuse and the importance of getting sober. The video will be followed by a 30-minute group discussion via zoom.
  Interventions: Behavioral: Education-only control group

INTERVENTIONS:
Behavioral: PST-APPLE Watch group — PST combined APPLE Watch is a tailored behavioral intervention that enables college students with AUD to successfully manage and overcome everyday life challenges influencing their alcohol intake and teach problem-solving skills.
  Arms: Treatment group
Behavioral: Education-only control group — Education-only control group receives Quit Drinking Motivation 20-min video created by the MotivationHub, followed by a 30-minute group discussion.
  Arms: Control group

SUMMARY:
The goals of this Pilot Trial are to test the preliminary efficacy of Problom-Solving Therapy (PST)-APPLE Watch in a 2-arm pilot Randomized Control Trial (RCT), vs education only-control to reduce alcohol use disorder symptoms and improve alcohol abstinence.

DETAILED DESCRIPTION:
The aims of this study are (1) to test feasibility & acceptability of screening for AUD symptoms/alcohol misuse and recruitment among college students, and (2) to test preliminary efficacy of PST-APPLE Watch in a 2-arm pilot Randomized Control Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Male and female college students aged 18-25 yr
* English-speaking
* Current alcohol use more than or equal to 2 days/week via phone screening
* Completion of AUDIT screening and meet criteria for (past year) mild, moderate or severe AUD during AUDADIS-5 interview
* Completion of written informed consent
* Interested in cutting back alcohol intake or changing his/her drinking
* Baseline screening study visit

Exclusion Criteria:

* Participation in past 6 months in AUD or substance use treatment
* Current use of medications used to treat AUD (e.g., naltrexone)
* Lifetime Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
* Current use of psychoactive drugs
* Not currently enrolled in college
* Not interested in cutting back alcohol intake or changing his/her drinking
* Pregnancy or intention to become pregnant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Alcohol abstinence | Up to 3 months
  Participants will be monitored for 3 months to assess alcohol abstinence by blood alcohol content.

SECONDARY OUTCOMES:
Change in AUD severity at 3 months. | Baseline, 3 months.
  Measured by Alcohol Use Disorder and Associated Disabilities Interview Schedule-5(AUDADIS-5). Change in AUD severity from baseline to 3 months.
Change in AUD frequency status. | Baseline, 3 months.
  Measured by AUDIT. Participants will be monitored for up to 3 months. This is the number of participants who screen positive for AUD.
Change in Alcohol-related negative consequences at 3 months. | Baseline, 3 months.
  Measured by Rutgers Alcohol Problem Index (RAPI).
Change in Alcohol use at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).
Change in Reasons for drinking at 3 months. | Baseline, 3 months
  Measured by Drinking Motives Questionnaire Revised (DMQ-R).
Change in negative affect at 3 months. | Baseline, 3 months
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in positive affect at 3 months. | Baseline, 3 months.
  Measured by Positive and Negative Affect Schedule (PANAS).
Change in Cognitive performance (executive cognitive ability and attention and working memory) at 3 months. | Baseline, 3 months.
  Compensatory Measured by Compensatory Cognitive Strategies Scale
Change in the quality of life at 3 months. | Baseline, 3 months.
  Measured by Quality of Life Scale (QOLS).
Percent heavy drinking days at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).
Percent binge drinking days at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).
Percent days abstinence at 3 months. | Baseline, 3 months.
  Measured by 90-day Timeline Followback (TLFB).

OTHER OUTCOMES:
Intervention Acceptability | 3 months.
  Measured by the Client Counseling Satisfaction Scale(CCSS).
Intervention Fidelity | 3 months.
  Participant adherence to the PST-APPLE intervention schedule will be assessed by documented session attendance.
Participant Retention | 3 months.
  Participant retention will be assessed throughout the study by monitoring the proportion of the sample retained at 3-month.
Protocol Acceptability | 3 months.
  PI or a trained research team member will conduct semi-structured interviews 3-month post-intervention with each participant and will adapt the semi-structured interview guide approach from the previous research study (Study named: Study of a PST-Trained Voice-Enabled Artificial Intelligence Counselor [SPEAC] and DEDICATE study).

CONTACTS AND LOCATIONS:
Overall Officials: Hallihan Hagar, PhD, RN, Principal Investigator — Department of Medicine, University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to the University of Illinois Chicago (UIC) Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of UIC Research Grants. Data from this research will be shared and the results of this research will be made available via publication in scientific journals and through scientific meetings where our findings are reported. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with typical scientific practices. All publications will be made publicly available consistent with UIC policies.
Supporting Information: SAP, CSR
Time Frame: After analyzing.